CLINICAL TRIAL: NCT01166867
Title: Photo-plethysmographic (PPG) Camera to Monitor Heart Rate, Respiration Rate and Oxygen Saturation in Infants.
Brief Title: A Pilot Study Using Photo-plethysmographic (PPG) Camera
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Children's Hospital of Orange County (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Willem Verkruysse, Ph.D., Associate Specialist, University of California, Irvine
Other Study IDs: 20097046
Record Dates: First submitted 2010-07-20; First posted 2010-07-21 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Infant Development
Keywords: assessment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infant Development: Photo-plethysmography monitoring
  Interventions: Device: Photo-plethysmography monitoring

INTERVENTIONS:
Device: Photo-plethysmography monitoring — monitoring vital sign in infant

SUMMARY:
The researcher want to use video signals to monitor heart rate, respiration rate and oxygen saturation using Photo-plethysmography (PPG) as the underlying mechanism for the method: periodic changes in skin reflectance, induced by the cardio-vascular wave, are measured using light.

DETAILED DESCRIPTION:
The Researcher want to use ambient light to monitor heart rate, respiration rate and oxygen saturation (SpO2) in infant patients in a hospital setting. The plethysmographic signal is typically strong on children. This provides a reliable heart rate monitor. However, to measure oxygen saturation, a quantitative value of the strength at two wavelength regions (green and red) is required. It is also not known if the normal ambient light is spectrally appropriate to analyze the video signals for oxygenation. With the current prototype of our system, we can monitor heart rate reliably and estimate oxygen saturation in adults, using normal artificial light or daylight, entering through a window.

ELIGIBILITY:
Inclusion Criteria:

* infant and toddler

Exclusion Criteria:

* non-infant

Ages: 1 Minute to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: infant
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Nelson, M.D, PhD, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (1):
- Children's Hospital of Orange County, Orange, California, United States